CLINICAL TRIAL: NCT03723564
Title: Serial Amnioinfusions as Regenerative Therapy for Pulmonary Hypoplasia in Fetuses With Intrauterine Renal Failure or Severe Renal Anomalies- a Feasibility Study
Brief Title: Serial Amnioinfusions as Regenerative Therapy for Pulmonary Hypoplasia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mauro H. Schenone, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-007726
Record Dates: First submitted 2018-10-02; First posted 2018-10-29 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Renal Failure Congenital; Congenital Renal Anomaly Nos; Renal Agenesis and Dysgenesis; Lower Urinary Tract Obstructive Syndrome
Keywords: bilateral renal agenesis; lower urinary tract obstruction; congenital renal anomalies; fetal surgery; amnioinfusion; fetus
MeSH Terms: conditions — Hereditary renal agenesis; Congenital Abnormalities | interventions — Ringer's Lactate; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Amnioinfusion (Experimental): Lactated Ringers Solution for Injection --- Serial ultrasound-guided amnioinfusion procedures will be performed on fetuses having severe LUTO or bilateral renal agenesis that are diagnosed between 18 0/7-25 6/7 weeks.
  Interventions: Drug: Lactated Ringers Solution for Injection

INTERVENTIONS:
Drug: Lactated Ringers Solution for Injection — Using ultrasound guidance, a 22 gauge needle will be introduced into amniotic cavity. Warmed Lactated Ringers solution will be injected into the amniotic cavity until an AFI of 8.0 cm is achieved
  Other Names: Lactated Ringers Solution for Infusion

SUMMARY:
Congenital lower urinary tract obstruction (LUTO) is a heterogeneous group of congenital anomalies that lead bladder outlet obstruction. If a complete obstruction is present, the perinatal mortality is estimated to be as high as 90% because of severe pulmonary hypoplasia due to the lack of amniotic fluid. Survivors have significant risk of renal impairment (90%) requiring dialysis or renal transplantation if no fetal intervention is performed.

Renal agenesis is the congenital absence of one or both kidneys due to complete failure of the kidney to form. As many as 33% of fetuses with bilateral renal agenesis are stillborn, and the rest of them die immediately after birth due to severe pulmonary hypoplasia.

The objective of the serial amnioinfusions for fetuses with these conditions will be to reduce the severity of pulmonary hypoplasia (regenerating the lung functionality) and therefore increase the chance that the newborn survives to begin peritoneal dialysis. Although there is initial evidence that serial amnioinfusions are feasible for the pregnant women and the fetuses, there is still a need to have a prospective clinical trial to confirm the hypothesis that serial amnioinfusions could prevent severe pulmonary hypoplasia allowing the newborns with bilateral renal agenesis or severe LUTO to survive to begin peritoneal dialysis.

Therefore, the investigators aim to study the hypothesis that serial amnioinfusions for fetuses with severe LUTO and renal failure and those with bilateral renal agenesis will reduce the severity of pulmonary hypoplasia and therefore increase the chance that the newborn survives to begin peritoneal dialysis.

DETAILED DESCRIPTION:
All women with fetuses having either severe LUTO with intrauterine renal failure or bilateral renal agenesis that meet the inclusion criteria will be invited to participate in this study. For those patients, the actual standard of care is expectant prenatal management or termination of pregnancy (<22 weeks according to law). This study will offer serial amnioinfusions for patients with LUTO or bilateral renal agenesis. Due to the rarity and complexity of these cases, the investigators expect to enroll a maximum of 5 women with affected fetuses per year. After two years (approximately 10 cases), a review of the data will be completed including all outcomes to determine whether to continue towards the original goal of treating 40 patients (20 mothers with affected fetuses) or to close the study,.

All procedures are anticipated to take place in the Family Birth Center at Mayo Clinic, Rochester. Serial ultrasound-guided amnioinfusion procedures will be performed on fetuses having severe LUTO or bilateral renal agenesis that are diagnosed between 18 0/7-25 6/7 weeks. This procedure will be performed in a sterile fashion within the operating room using the same technique that is routinely used to perform the ultrasound-guided amnioinfusion. Once consented, weekly ultrasound monitoring will be conducted and if the amniotic fluid index (AFI) is determined to be <2 cm, amnioinfusion will proceed. Prior to each infusion, 5mLs of amniotic fluid will be collected to study surrogate markers of lung function (research only). Using a 22-gauge needle, warm sterile lactated ringer solution will be infused into the amniotic cavity until the AFI is equal to 8 cm. Some studies have demonstrated that the composition of the amniotic fluid during second and third trimester is closer to the lactated ringer solution. This procedure will be continued weekly until the fetus reaches 34 weeks, after which only monitoring will occur. If preterm premature rupture of the membranes (PPROM) occurs prior to 34 weeks, no further amnioinfusion procedures will be performed. Patients with PPROM will be managed according to the standardized clinical management. The anticipated length of stay in the hospital after each infusion is approximately 2 days if no uterine contractions are observed.

The prenatal care, delivery and postnatal management of the infant will be conducted according to the standardized clinical care. Delivery will be scheduled at the Mayo Clinic Family Birth Center and the infants will be followed for 24 months by the multi-specialty team as part of the standard clinical management including follow-up with neonatologist (NICU team), pediatric nephrology and transplant team according to the clinical protocol for postnatal renal replacement therapy and transplant. Neurodevelopment of the children will assessed using a combination of clinical examination and the Bayley Scale of Infant Development during the first 24 months of life.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with singleton uterine pregnancy
* Maternal age > age 18
* Fetus < 26 weeks gestational age with severe LUTO and intrauterine renal failure
* Fetus < 26 weeks gestational age with bilateral renal agenesis
* Fetus with absence of chromosome abnormalities
* Fetus with absence of associated anomalies
* Mother has negative Hepatitis B, Hepatitis C, and HIV testing
* Mother meets psychosocial criteria that allows her to make a conscious decision about her fetus/infant

Exclusion Criteria:

* Associated fetal anomaly unrelated to LUTO or renal agenesis
* Increased risk for preterm labor including short cervical length, history of incompetent cervix with or without cerclage, and previous preterm birth
* Placental abnormalities known at time of enrollment
* Maternal-fetal Rh isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia affecting the current pregnancy
* Maternal medical condition that is a contraindication to surgery or anesthesia
* Mother has declined invasive testing
* Inability to comply with the travel and follow-up requirements of the trial
* Participation in another interventional study that influences maternal and fetal morbidity and mortality
* Participation in this clinical trial during a previous pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | First amnioinfusion through delivery which may be up to 22 weeks.
  Total number of Adverse Events experienced

SECONDARY OUTCOMES:
Survival to renal transplant | 5 years
  Number of subjects able to receive renal transplant.
Survival to dialysis | From time of birth up to one month
  Number of subjects able to receive dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Schenone, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials